CLINICAL TRIAL: NCT05352776
Title: Sensing and Defibrillation With a Commercially Available ICD Coupled With a Parasternal Extravascular Lead (SECURE EV) Study
Acronym: SECURE EV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AtaCor Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: DOC-10181
Record Dates: First submitted 2022-04-22; First posted 2022-04-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Ventricular Arrhythmia; Ventricular Tachycardia; Ventricular Fibrillation
Keywords: Ventricular Defibrillation; Extravascular
MeSH Terms: conditions — Tachycardia, Ventricular; Ventricular Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AtaCor EV-ICD Lead System (Experimental): Subjects implanted with the AtaCor EV-ICD Lead Model AC-7001
  Interventions: Device: AtaCor EV-ICD Lead

INTERVENTIONS:
Device: AtaCor EV-ICD Lead — Subjects will receive the AtaCor EV-ICD Lead being evaluated in the study.

SUMMARY:
The SECURE EV Study is a prospective, multi-center, single-arm study without concurrent or historical controls. The objectives of the study are 1) to characterize safety of the AtaCor EV-ICD Lead up to 90 days post-implant, and 2) to characterize sensing and conversion of induced VF up to 90 days post-implant.

DETAILED DESCRIPTION:
The primary safety objective of the study is to characterize safety of the AtaCor EV-ICD Lead up to 90 days post-implant. The primary performance objective is to characterize sensing and conversion of induced VF up to 90 days post-implant.

Up to 3 Investigational Sites Worldwide will participate with up to 20 subjects enrolled in the study. Patients undergoing de novo or replacement ICD procedure will be eligible for participation. Study participation requires sub-chronic evaluation of the lead up to 90 days.

Subjects will receive a concomitant EV-ICD System, comprising the investigational EV-ICD Lead connected to a commercially available ICD. Prior to discharge, the EV-ICD will be programmed to monitor only to detect and store ventricular arrhythmias over the 90-day follow-up period.

After the EV-ICD System is removed (up to 90 days post-implant), the Subject will be followed for an additional 30 days then exit the study. The duration of study participation for an individual Subject is 120 ± 7 days. The study is expected to complete within 6 months of the first enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old
2. Indicated for de novo or replacement ICD procedure

Exclusion Criteria:

1. NYHA IV functional class
2. BMI ≥ 35 kg/m2
3. Inotropic therapy in past 180 days
4. Subjects who require continual ventricular pacing
5. Presence or planned use of a subcutaneous ICD lead, subcutaneous coils/arrays, epicardial patches or epicardial pace/sense leads within the study period.
6. Planned MRI within the study period
7. Subjects on anticoagulation or antiplatelet therapy that cannot be temporarily discontinued for the procedure
8. Logistical or safety related circumstances that may prevent data collection or follow-up
9. Participation in any concurrent clinical study without prior written approval from the Sponsor
10. Inability to give an informed consent to participate in the Study

    Known prior history for any of the following:
11. Structural abnormalities of the heart that may increase risk of the study procedure or an obstructed/restricted pathway into the mediastinum for the EV-ICD Dilator, EV-ICD Delivery Tool and EV-ICD Lead
12. Uncontrolled paroxysmal, persistent or permanent atrial fibrillation
13. Median or partial sternotomy
14. Surgery with disruption of the lung, pericardium or connective tissue between the sternum and pericardium
15. Significant anatomic derangement of or within the thorax (e.g., pectus excavatum, significant scoliosis)
16. Thoracic radiation therapy, pneumothorax, pneumomediastinum or other medical treatments/conditions which may complicate the EV-ICD Lead insertion procedure
17. Pericardial disease, pericarditis and mediastinitis
18. Medical treatments, surgeries or conditions that increase the potential for pericardial adhesions
19. FEV1 < 1.0 Liter
20. Surgically corrected congenital heart disease (not including catheter-based procedures)
21. Allergies to the device materials as listed in the Instructions for Use (IFU)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Incidence of ADEs | Up to 120 days post-implant
  Incidence of Adverse Device Effects (ADEs)
Induced VF Conversion Success | Up to 90 days post-implant
  Induced VF conversion success with ≥10 J safety margin 60-90 days post-implant

SECONDARY OUTCOMES:
Lowest Defibrillation Conversion Energy | Procedure
  Lowest Defibrillation Conversion Energy (J) at implant with left mid-axillary PG location
Induced VF Conversion Success - Implant | Procedure
  Induced VF conversion success rate at implant with left pectoral PG location
Induced VF Conversion Success - 30 Days | Up to 30 days post-implant
  Induced VF conversion success with ≥10 J safety margin at 30 days
Sensing and Detection of Ventricular Arrhythmias | Up to 90 days post-implant
  Ability to automatically sense and detect induced and spontaneous ventricular arrhythmias
Detection Time for VT/VF | Up to 90 days post-implant
  Detection time for spontaneous VT/VF episodes recorded during follow-up by the permanent TV-ICD System and concomitantly implanted investigational EV-ICD System
Detection Time and Time-to-Therapy | Up to 90 days post-implant
  EV-ICD VF detection time and time-to-therapy
Brady Pacing Electrical Performance: Pacing Capture Threshold | Up to 90 days post-implant
  Pacing Capture Threshold (V)
Brady Pacing Electrical Performance: Pacing Impedance | Up to 90 days post-implant
  Pacing Impedance (ohms)
Brady Pacing Electrical Performance: R-wave Amplitude | Up to 90 days post-implant
  R-wave Amplitude (mV)

CONTACTS AND LOCATIONS:
Overall Officials: Martin C Burke, DO, Principal Investigator — AtaCor Medical, Inc.
Locations (1):
- Sanatorio Italiano, Asunción, Paraguay

IPD SHARING:
Plan to Share IPD: No